CLINICAL TRIAL: NCT05486299
Title: Clinical Study of the Safety of a Single-port Endoscopic Surgical System for General Surgery: An Exploratory Study of a Novel Robotic System
Brief Title: Clinical Study of the Safety of a Single-port Endoscopic Surgical System for General Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Director, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RASIS-01
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: General Surgery
Keywords: robotic surgery; robotic assisted single-incision surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-port Endoscopic Surgical System (Experimental): A novel robotic surgical system that can be configured for multi-port, single-port, or hybrid-port procedures. In the single-port configuration, a four-channel trocar shall be used. The surgical tools are steered through the curved access channels in the trocar to enter a patient's abdomen.
  Interventions: Procedure: Robotic assisted single-port general surgery

INTERVENTIONS:
Procedure: Robotic assisted single-port general surgery — Robot assisted single-port rectal resection, colectomy, partial gastrectomy, appendectomy and cholecystectomy via the single-port configuration

SUMMARY:
This is a small-scale pre-clinical exploratory study to investigate the safety of a novel single-port robotic system for general surgery.

DETAILED DESCRIPTION:
Single-incision laparoscopic surgery is a surgical procedure in which multiple laparoscopic instruments are placed through a single small incision. It has the advantages of less surgical trauma, better cosmetic results and less postoperative pain compared with conventional laparoscopic surgery. However, the technical challenges and difficulties, including loss of triangulation, parallel coaxial effect, difficulty of achieving correct exposure, shared fulcrum, lack of ergonomic favorable position, etc. limited its widespread use. Robot-assisted laparoscopic surgery have significant advantages such as minimally invasive, delicate, and flexible, which can greatly expand the surgeon's surgical capabilities and effectively solve the various problems faced by traditional surgery. Therefore, robotic assisted single-port surgery is attracting increasing attention. This study is to investigate the safety of a novel single-port robotic system for general surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age ≤75 years
* Suitable for minimally invasive surgery
* 18.5≤BMI≤28 kg/m2
* ASA score is Ⅰ-Ⅲ
* Informed consent
* Colon and rectal resection: colon and rectal polyps, inflammatory bowel disease, intestinal diverticula, colorectal cancer diagnosed cT3N0M0 with a maximum diameter of ≤4 cm located above the peritoneal reflection.
* Partial gastrectomy: gastric stromal tumor, gastric giant ulcer.
* Appendectomy: chronic appendicitis.
* Cholecystectomy: chronic cholecystitis combined with gallbladder stones, gallbladder polyps (> 1 cm).

Exclusion Criteria:

* With other malignancies or a previous history of other malignancies
* Undergone other major surgical treatment within 3 months prior to enrolment or planned during the trial
* With active tuberculosis
* With severe systemic disease
* With long-term use of anticoagulant and anti-platelet drugs (anti-platelet aggregation drugs discontinued less than 1 week prior to surgery), history of bleeding disorders or hematopoietic or coagulation disorders.
* With severe allergies and suspected or established alcohol, drug or substance addiction
* Patients who are immunodeficiency virus (HIV) antibody positive; hepatitis B surface antigen (HbsAg) positive and have a hepatitis B virus DNA (HBV-DNA) copy number above the lower limit of detection or normal range; hepatitis C virus (HCV) antibody positive; syphilis spirochete antibody positive and at high risk of transmission as judged by the investigator.
* Emergency surgery
* Women who are pregnant, breastfeeding or planning to become pregnant during the trial
* Other conditions which, in the opinion of the investigator, make participation in this trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | intraoperative
  The proportion of converted to laparotomy, laparoscopic surgery and added ≥ 2 trocars

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Length of stay | 1-14 days after surgery
  The postoperative day when patients complied with the predefined discharge criteria（days after surgery）
Early morbidity rate | 30 days after surgery
  morbidity rate 30 days after surgery
Incision healing | 1-14 days after surgery
  Incision healing grade at discharge. Grade A: well healed; Grade B: incision with inflammatory reaction but no suppuration; Grade C: incision cracked and suppurating

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, MD, PHD, Study Chair — Ruijin Hospitlal , Shanghai Jiaotong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grochola LF, Soll C, Zehnder A, Wyss R, Herzog P, Breitenstein S. Robot-assisted versus laparoscopic single-incision cholecystectomy: results of a randomized controlled trial. Surg Endosc. 2019 May;33(5):1482-1490. doi: 10.1007/s00464-018-6430-7. Epub 2018 Sep 14. PMID 30218263
- [Background] Lim MS, Melich G, Min BS. Robotic single-incision anterior resection for sigmoid colon cancer: access port creation and operative technique. Surg Endosc. 2013 Mar;27(3):1021. doi: 10.1007/s00464-012-2549-0. Epub 2012 Oct 10. PMID 23052525
- [Derived] Guo Z, Shi Y, Song Z, Jia W, Wang S, Zhang Y, Ji X, Liu K, Zhang T, Cheng X, Zhao R. Single-incision robotic assisted surgery: a nonrandomized cohort pilot study on a novel surgical platform in colorectal surgery. Int J Surg. 2023 Nov 1;109(11):3417-3429. doi: 10.1097/JS9.0000000000000612. PMID 37526117